CLINICAL TRIAL: NCT01740440
Title: Effect of a Transcutaneous Electrical Nerve Stimulation (TENS) Device on Overall Facial Appearance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bio-Medical Research, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SRG-BMR Face01
Record Dates: First submitted 2012-11-21; First posted 2012-12-04 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Ageing
Keywords: Healthy females

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMR Face treatment (Other): BMR Face treatment used once a day for 12 weeks
  Interventions: Device: BMR Face

INTERVENTIONS:
Device: BMR Face — BMR Face used in accordance with manufacturer IFU

SUMMARY:
Safety and clinical performance of the BMR Face device (manufactured by Bio-Medical Research)

DETAILED DESCRIPTION:
Evaluate the efficacy of the BMR Face device in relation to facial appearance at 12 weeks compared to baseline. Efficacy will be assessed by overall facial improvement assessed live by the Investigator and a subject assessment of facial appearance including the Global Aesthetic Improvement Scale (GAIS).

The Global Aesthetic Improvement Scale is a five-grade subjective test. The physician and patient independently describe the degree of improvement in facial appearance. Possible responses were (1) Significantly marked improvement, (2) marked improvement, (3) moderate improvement, (4) slight improvement, (5) no improvement

Secondary objectives are to evaluate safety and further evaluate the subject's and investigator's satisfaction (both a live and blinded assessor) with the BMR Face treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPAA authorization
* Subjects who are healthy females between 35 and 55 years of age
* Subjects with a Body Mass Index (BMI) between 15-35 kg/m2 (light underweighted to light obese)
* Subjects may have all skin types
* Subjects with age related skin laxity in the treatment area
* Subjects who agree not to have any procedures affecting facial volume (any fillers or fat transfer) for the duration of the study
* Subjects who agree not to have any other procedures affecting skin quality (microdermabrasion, resurfacing, peels, lasers, acne treatments, etc.) for the duration of the study
* Subjects who agree to make no changes in their existing skincare regime during the study period
* Subjects who agree to avoid excessive sun radiation or use appropriate sun protection with SPF 30 or higher
* Subjects who agree not to alter their diet for the duration of the study
* Subjects who understand this study and are able to follow study instructions and are willing to attend the required study visits
* Subjects who agree to be photographed for the purposes of the study and give consent for these photographs to be used in marketing advertisements where their identity will not be concealed in these photographs

Exclusion Criteria:

* Subjects who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy.
* Subjects of child-bearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence)
* Subjects who cannot understand or are not willing to comply with the requirements of the study
* Subjects who have any dermatologic conditions including acne, rosacea, eczema, psoriasis, severe sun damage or scars within the treatment area
* Subjects who have any known cancer including skin cancers (Basal Cell Carcinoma, Squamous Cell Carcinoma and Melanoma)
* Subjects with a history of heart disease or stroke
* Subjects who have any active implanted medical devices (pacemaker, pump etc)
* Subjects having any metal implants. Dental implants and fillings are allowed as well as piercings as long as they are not in the treatment area.
* Subjects who have used a tanning bed in the past four weeks or plan to use a tanning bed for the duration of the study
* Subjects who are HIV positive
* Subjects who have had systemic corticosteroid therapy in the past 6 months
* Subjects who have had a facial dermabrasion, chemical peel, laser, or IPL treatment in the past 6 months
* Subjects who have used botulinum toxin, hyaluronic acid, collagen, fat injections and /or other methods of skin augmentation (enhancement with injected or implanted material) in the past 6 months
* Subjects who have had ablative resurfacing procedure, brow lift, blepharoplasty or face lift in treated area in the past 12 months
* Subjects who have had any other surgery in treated area in the past 12 months
* Subjects who have an existing medical condition that the Investigator considers may put the subject at risk or compromise their participation in the study
* Subjects who have participated in another research study in the past 30 days
* Subjects who are currently involved in any injury litigation claims
* Subjects who have used the BMR Face device previously

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sadick, Dr, Principal Investigator — Sadick Research Group
Locations (1):
- Sadick Research Group, New York, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BMR Face Treatment: BMR Face treatment used once a day for 12 weeks
  BMR Face
Period: Overall Study
Arm/Group | BMR Face Treatment
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | BMR Face Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (3.7)
Sex/Gender, Customized [Number; unit: female participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Overall Facial Improvement Assessed Live by the Investigator and Subjects Using the Global Aesthetic Improvement Scale (GAIS) at 12 Weeks Compared to Baseline.
Description: Evaluate the efficacy of the Efficacy will be assessed by overall facial improvement assessed live by the Investigator and a subject assessment of facial appearance including the Global Aesthetic Improvement Scale (GAIS).
  The Global Aesthetic Improvement Scale is a five-grade subjective test. The physician and patient independently describe the degree of improvement in facial appearance. Possible responses were (1) Significantly marked improvement, (2) marked improvement, (3) moderate improvement, (4) slight improvement, (5) no improvement.
  For reporting of outcomes, the higher the GAIS value, the greater the improvement (Range 0-4).
Time Frame: 12 weeks
Population: 23 out of 30 subjects that were enrolled in the study were statistically analyzed. 3 subjects were lost to follow-up and 4 subjects had to be excluded from analysis due to protocol violations.
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | BMR Face Treatment
Number analyzed (Participants) | 23
Scores on a Scale
  GAIS (Investigator) | 2.17 [0 to 4]
  GAIS (Subject) | 2.26 [0 to 4]

2. Secondary Outcome: To Evaluate Overall Facial Improvement Assessed Live by the Investigator and Subjects Including the Global Aesthetic Improvement Scale (GAIS) at 6 Weeks Compared to Baseline
Description: as for outcome 1
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BMR Face Treatment
Number analyzed (Participants) | 23
units on a scale
  GAIS (Investigator) | 2.04 [0 to 4]
  GAIS (Subject) | 1.26 [0 to 4]

3. Secondary Outcome: To Evaluate the Subject's Satisfaction With BMR Face Treatment at 6 Weeks and 12 Weeks (Subject Self- Assessment).
Description: The Subject Satisfaction Assessment Scale is a 5 point scale where a subject rates their satisfaction level as Very Satisfied, Satisfied, No Opinion, Unsatisfied or Very Unsatisfied.
Time Frame: 6 weeks, 12 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | BMR Face Treatment
Number analyzed (Participants) | 23
percentage of subjects
  Week 12 - Very Satisfied | 34.8
  Week 12 - Satisfied | 47.8
  Week 12 - No opinion | 4.3
  Week 12 - Unsatisfied | 13.0
  Week 6 - Very Satisfied | 17.4
  Week 6 - Satisfied | 39.1
  Week 6 - No opinion | 30.4
  Week 6 - Unsatisfied | 13.0

ADVERSE EVENTS:
Time Frame: Subject were followed for Adverse Events for the duration of their participation in the study (up to 12 weeks)
Arm/Group | BMR Face Treatment
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other